CLINICAL TRIAL: NCT01548014
Title: Reduction in Frequency of Infliximab Administration From q 8 Weeks to q 12 Weeks in Children With Crohn's Disease Receiving Probiotic VSL#3 Supplementation: A Pilot Study
Brief Title: The Effect of a Probiotic Preparation (VSL#3) Plus Infliximab in Children With Crohn's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, YonHo Choe, Pediatrics, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009-11-046
Record Dates: First submitted 2012-02-17; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; VSL #3; infliximab
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: VSL#3 — children with severe Crohn's disease were assigned in a 1:1 ratio with either IFX 5 mg/kg q 12 weeks + concurrent immunomodulator + VSL#3 (4 sachets of 450 x 109 organisms per day) (Group A), or IFX 5 mg/kg q 8 weeks + concurrent immunomodulator (Group B).
  Other Names: VSL#3 : the living shield(probiotics)

SUMMARY:
The purpose was to evaluate as to whether administration of infliximab of 12 week interval with supplementary VSL#3 is more effective or at least of similar efficacy when compared to conventional administration of infliximab only of 8 week interval.

DETAILED DESCRIPTION:
The purpose of our study was to evaluate if supplementation of VSL#3 can improve treatment outcome for those pediatric Crohn's patients treated with infliximab every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who were diagnosed with severe Crohn's disease who require infliximab treatment
* confirmed diagnostic of Crohn's disease in clinical, endoscopic and histological findings

Exclusion Criteria:

* patients who has proven to have infliximab antibody

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-09 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Frequency of Infliximab Administration from q 8 Weeks to q 12 Weeks in Children with Crohn's Disease Receiving Probiotic VSL#3 Supplementation | 1-year treatment period
  Disease Activity Index (PCDAI) scores, hematocrit, albumin, ESR, CRP, TNF-α, IL-8, INF-γ, and endoscopic findings (Simple Endoscopic Score for Crohn's Disease was used) were assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea